CLINICAL TRIAL: NCT00429650
Title: Using the Energy Gap to Prevent Weight Regain
Acronym: Lose-It
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 06-0369; R01DK071692 (NIH)
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Obesity
Keywords: Weight maintenance; Weight loss
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Increased amount of exercise to maintain weight loss.
  Interventions: Behavioral: increased exercise
- 2 (Experimental): Combination of Exercise and Diet to maintain weight loss
  Interventions: Behavioral: Exercise and Diet
- 3 (Active Comparator): Use diet alone to maintain weight loss.
  Interventions: Behavioral: diet

INTERVENTIONS:
Behavioral: increased exercise — Use prescribed number of minutes of exercise 5-6 days per week to maintain weight loss.
  Arms: 1
Behavioral: diet — Use a prescribed diet to maintain weight loss
  Arms: 3
Behavioral: Exercise and Diet — Use a combination of exercise and diet to maintain weight loss.
  Arms: 2

SUMMARY:
The major challenge in obesity treatment is not producing weight loss but in preventing that weight from being regained. There are many different methods to lose weight, but there are no recommendations for how you can best achieve long-term weight loss maintenance. Despite the method used to reduce one's body weight, very few of these individuals are able to keep their weight off permanently. This project aims to identify how much activity is necessary to prevent weight regain after weight loss.

ELIGIBILITY:
Inclusion Criteria:

1. All ethnic groups and both genders
2. Age: Lower age limit: 19 years; Upper age limit: 45 years
3. Body-mass Index: Lower BMI limit: 30 kg/m2; Upper BMI limit: 40 kg/m2 and weight stable within +/- 5 pounds in the last 6 months, and currently at maximum non pregnant body weight (+/- 5%)
4. A negative treadmill stress test or subsequent follow up cardiac testing for cardiac ischemia.

Exclusion Criteria:

1. History of cardiovascular disease, including coronary artery disease, congestive heart failure, & unstable angina, or uncontrolled hypertension ( > 140/90 mm Hg)
2. Currently smoking or stopped smoking in the last 12 months
3. Medications affecting weight, energy intake, or energy expenditure in the last 6 months
4. Use of oral steroids within the last 12 months
5. History of stroke or seizures, thyroid disease, type 1 or 2 diabetes, Cushings syndrome, cerebrovascular, renal disease, hepatic disease, arrhythmias
6. Cancer requiring treatment in the past 5 years, with the exception of skin cancers other than melanoma
7. Infectious diseases: Self-reported HIV positivity or Active tuberculosis
8. Weight loss or weight gain of > 5% in past 6 months for any reason except post-partum weight loss
9. Likely to move away in next 1.5 years
10. Inability to adhere to the program such as inability to increase walking
11. Currently pregnant, lactating or less than 6 months post-partum
12. Major psychiatric disorder: Exclusions related to medications -Antipsychotic agents (these include, but are not limited to: Haldol, Loxitane, Mellaril, Navane, Prolixin, Stelazine, Thorazine, and Trilafon)
13. Current depression by history or Beck Depression Inventory (BDI)
14. Currently being treated for psychological condition

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 175 (Actual)
Dates: Start 2007-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in Weight | 18 Months

CONTACTS AND LOCATIONS:
Overall Officials: Holly R. Wyatt, MD, Principal Investigator — University of Colorado at Denver Health Sciences Center
Locations (1):
- Center for Human Nutrition, Denver, Colorado, United States

REFERENCES:
- [Derived] Polsky S, Garratt Ogden L, Scown Maclean P, Danielle Giles E, Brill C, Roxanna Wyatt H. Biomarker Profile Does Not Predict Weight Loss Success in Successful and Unsuccessful Diet-Reduced Obese Individuals: a Prospective Study. ISRN Obes. 2013 Jan 1;2013:804129. doi: 10.1155/2013/804129. PMID 24363955